CLINICAL TRIAL: NCT04520191
Title: Home-based Kidney Care in Native Americans of New Mexico (HBKC) - COVID-19 Related Disruption in Health and Health Care
Brief Title: Home-based Kidney Care in Native Americans of New Mexico (HBKC) - Enhancement: COVID-19 Study
Status: Completed | Type: Observational
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Vallabh O Shah, Professor, University of New Mexico
Other Study IDs: 16-344-Enhancement
Record Dates: First submitted 2020-08-17; First posted 2020-08-20 (Actual); Results first posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: CKD
Keywords: CKD, Diabetes, Ameircan Indians, COVID-19,
MeSH Terms: conditions — Diabetes Mellitus; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Novel severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) OR COVID-19 related Addition: The aim of this addition activity is to track the impact of the COVID-19 epidemic on participants with diabetes and chronic kidney disease (CKD). Investigators have modified the original HBKC Study protocol to expand data currently collected from study participants to include data in the following domains linked to the COVID-19 epidemic:

symptoms of COVID-19 disease, access to healthcare, and impact on health related behaviors (such as medication adherence, physical activity, dietary behaviors, smoking, and alcohol use).

DETAILED DESCRIPTION:
Investigators will administer a survey by phone or mail to all participants screened for diabetes and chronic kidney disease in the original HBKC study protocol. The survey will address to the following aims:

Aim 1. Develop a phone-based and or mail based survey to understand the impact of COVID19 on patient-reported outcomes for adults with diabetes and CKD.

Aim 2. Test the feasibility and acceptability of this phone-based and or mail based survey in the HBKC cohort.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate in the phone-based and or mail based survey.

Exclusion Criteria:

* None

Ages: 21 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All Native Americans (n=529) who participated in the screening for diabetes and kidney disease as part of original HBKC study will be approached for this survey based study.
Sampling Method: Non-Probability Sample
Enrollment: 309 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited 309 participants from 540 individuals who were initially approached by phone and/or mailings from September 2020 to July 2021 to participate in the survey.
Groups:
- Covid Survey: COVID-19 Survey.
Period: Overall Study
Arm/Group | Covid Survey
Started | 309
Completed | 309
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Single Group Survey: Survey of the entire group
Arm/Group | Single Group Survey
Number analyzed (Participants) | 309
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 197
  Male | 112
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 309
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Problems in Their Health Care Due to COVID-19 Related Isolation
Description: Document COVID-19 disruptions in normal health care check-ups, transportation, economic status, and access to food and water.
Time Frame: six months
Measure: Count of Participants; unit: Participants
Groups:
- COVID Survey: COVID Survey
Arm/Group | COVID Survey
Number analyzed (Participants) | 309
Participants | 155

ADVERSE EVENTS:
Time Frame: 6 months
Description: This is a survey of minimum risk.
Groups:
- Single Group Survey: Single Group Survey
Arm/Group | Single Group Survey
All-Cause Mortality (participants affected / at risk) | 0/309
Serious Adverse Events (participants affected / at risk) | 0/309
Other Adverse Events (participants affected / at risk) | 0/309

LIMITATIONS AND CAVEATS:
Participant selection bias. The survey instruments have not been fully validated for American Indians.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2021-05-13): https://cdn.clinicaltrials.gov/large-docs/91/NCT04520191/Prot_000.pdf